CLINICAL TRIAL: NCT06479850
Title: A Strength-Based Intervention to Improve Job Interview Skills in Neurodiverse Young Adults
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kessler Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: E-1251-24
Record Dates: First submitted 2024-06-17; First posted 2024-06-28 (Actual); Last update posted 2024-07-24 (Actual); Status verified 2024-07

CONDITIONS: ADHD; Dyslexia; Learning Disabilities
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Dyslexia; Learning Disabilities | interventions — Gene Expression

STUDY DESIGN:
Intervention Model Description: Kessler Foundation Strength Identification and Expression (KF-STRIDE®
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment Group (Experimental): In this arm, participants would participate in in an intervention program that uses character strengths to improve job maintenance skills in young adults.
  Interventions: Behavioral: KF-STRIDE®
- Control Group (No Intervention): In this arm, participants are services as usual and will participate in their regular activities.

INTERVENTIONS:
Behavioral: KF-STRIDE® — Treatment group will receive 12 web based sessions of a strength-based training tool (once or twice a week). Sessions are approximately 60 minutes long.
  Other Names: Kessler Foundation Strength Identification and Expression
  Arms: Treatment Group

SUMMARY:
the investigators are looking to evaluate the effectiveness of a strength-based program in improving job interview skills in neurodiverse young adults. This program is designed to help participants understand and speak to others about their personal qualities and abilities. The investigators are examining the effects of this program in young adults who may have difficulty with job interviews, and who may want to improve these skills. Some of these young adults have received special education services in the past for learning differences, such as attention deficit hyperactivity disorder (ADHD) or dyslexia.

DETAILED DESCRIPTION:
Practicing job interview skills has been identified as an important target for job employment services in N-TAY. However, the majority of studies using interventions in neurodiverse individuals have taken a deficit-based approach (i.e. to fix what is deficient in a person). This approach has triggered increasing criticism and dissatisfaction from the disability community. Further, focusing on deficits will not result in identification, awareness, or expression of strengths, important skills needed for self-advocacy and transition to adulthood. KF-STRIDE takes a strength-based approach, using principles of positive psychology to help N-TAY identify and express their unique character strengths to future employers. Over the course of a recently funded pilot study, the team has evaluated the efficacy of KF-STRIDE in those on the autism spectrum. The investigators have found that individuals on the spectrum who train with KF-STRIDE show improved job interview skills, and preliminary data indicates that they also have improved chances of obtaining employment in the community. However, KF-STRIDE has never been evaluated in youth other than those on the spectrum, including those with ADHD, dyslexia or other learning differences which may benefit from the training. The investigators aim to evaluate the preliminary effectiveness of KF-STRIDE in a randomized controlled trial comparing KF-STRIDE to services as usual (SAU) to improve employment, as well as identify mechanistic targets which may lead to improved employment, and to evaluate the fidelity, acceptability, usability, and feasibility of the proposed intervention, KF-STRIDE, via initial process evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Lives in the United States of America
* Between the ages of 14-26 Speaks English well
* At a 4th grade reading level

Exclusion Criteria:

* Had a stroke, Traumatic Brain Injury, or neurological injury or disease in the past(like brain tumor or epilepsy)
* Has a history of significant psychiatric illness(like schizophrenia or psychosis)
* Has uncontrolled seizures or other unstable medical complications

Ages: 14 Years to 26 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-08-01 (Estimated); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Mock Job Interview | [Time Frame: Baseline, Immediate Post-Test between weeks 7 and 8]
  Blinded reviewers using a standardized scoring measure will rate the video recorded mock job interviews, where the minimum total value is a 0 and the maximum total value is 77, with higher scores meaning a better outcome.
Employment Status | Baseline, Immediate Post-Test between weeks 7 and 8, and 6 months Post-Test
  We will examine whether the person became employed or other changes to their employment status. Yes=1, No=0
Time-to-reach Employment | 6 months Post-Test
  We will examine how long it took for the person to obtain employment. Assessed as weeks since intervention completion.
Strength Knowledge and Strengths Use Scale (SKUS) | Baseline, Immediate Post-test between weeks 7 and 8
  Measure to assess knowledge and use of one's strengths and measure changes following strengths-based interventions. Two scores: Strengths Use and Strengths Knowledge. Strengths Use values range from 14-98, with higher score indicating a better outcome. Strengths Knowledge values range from 8-56, with higher score indicating a better outcome
Youth Interview- Self Efficacy and Anxiety | Baseline, Immediate Post-test between weeks 7 and 8
  25 items combined, about confidence and interview comfort in adolescents, with values ranging from 0 to 5 for each item, and higher scores meaning a better outcome.
Job Search Behavior Scale | Baseline, Immediate Post-test between weeks 7 and 8
  12 items measuring how often one engages in job search activities- language modified for use in youth, with values ranging from 1-5, with higher scores meaning a better outcome.
Work Readiness Scale | Baseline, Immediate Post-test between weeks 7 and 8
  13 items about the perception of one's ability to work, with values ranging from 1 to 5, with higher scores meaning a better outcome.
Global Assessment of Character Strengths (GACS) | Baseline, Immediate Post-test between weeks 7 and 8
  24 items measuring one's identification of personal character strengths, with values ranging from 1 to 5, with higher scores meaning a better outcome

CONTACTS AND LOCATIONS:
Overall Officials: Helen Genova, Principal Investigator — Kessler Foundation

IPD SHARING:
Plan to Share IPD: No